CLINICAL TRIAL: NCT03715751
Title: Adaptive Support Ventilation in Acute Respiratory Distress Syndrome
Acronym: ARDS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Responsible Party: Principal Investigator, Daniel Talmor, Edward Lowenstein Professor of Anesthesia, Beth Israel Deaconess Medical Center
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 2017P000596
Record Dates: First submitted 2018-08-15; First posted 2018-10-23 (Actual); Last update posted 2022-03-08 (Actual); Status verified 2022-03

CONDITIONS: Acute Respiratory Distress Syndrome
Keywords: Adaptive Support Ventilation; ARDS; Esophageal Pressure; Mechanical Ventilation; Transpulmonary Pressure
MeSH Terms: conditions — Respiratory Distress Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ASV (Active Comparator): Patients in this arm will have the ventilator adjusted per results of recent arterial blood gas. Esophageal balloon placement will be confirmed. Study team will measure several tidal breaths, end-expiratory and end-inspiratory ventilator holds. Then PEEP will be adjusted to achieve desired end-expiratory transpulmonary pressures, Fraction of Inspired Oxygen (FiO2) adjusted as needed to achieve SpO2>95%, and Tidal Volume (Vt) adjusted to 6cc/kg (IBW). Respiratory Rate (RR) will be adjusted to target the same minute ventilation achieved prior to any change in Vt. Patients will then be switched to ASV mode. The percentage minute volume (%minVol) will be adjusted to target the same minute ventilation as was achieved before the change. Settings will be maintained for approximately 1-2 hours, after which breath hold measurements will be repeated and another blood gas drawn.
  Interventions: Other: ASV
- Lung Protective Ventilation (Active Comparator): Patients in this arm will have the ventilator adjusted per results of recent arterial blood gas. Esophageal balloon placement will be confirmed. Study team will measure several tidal breaths, end-expiratory and end-inspiratory ventilator holds. Then PEEP will be adjusted to achieve desired end-expiratory transpulmonary pressures, Fraction of Inspired Oxygen (FiO2) adjusted as needed to achieve SpO2>95%, and Tidal Volume (Vt) adjusted to 6cc/kg (IBW). Respiratory Rate (RR) will be adjusted (while leaving the Vt at 6cc/kg) to achieve the same minute ventilation. Patients will then be maintained on their current lung protective ventilation settings for approximately 1-2 hours, after which breath hold measurements will be repeated and another blood gas drawn.
  Interventions: Other: Lung Protective Ventilation

INTERVENTIONS:
Other: ASV — Adaptive Support Ventilation
  Other Names: Adaptive Support Ventilation
  Arms: ASV
Other: Lung Protective Ventilation — Targeted tidal volume of 6cc/Kg, Positive Inspiratory Pressure titrated per ARDS guidelines.
  Arms: Lung Protective Ventilation

SUMMARY:
The purpose of this protocol is to compare standard of care lung protective ventilation settings with an automated ventilator setting, called Adaptive Support Ventilation (ASV), in patients with acute respiratory distress syndrome (ARDS). This study will compare measurements (i.e. tidal volumes, driving pressure, respiratory rate (RR), compliance, peak airway pressures, plateau pressures, PEEP) with each ventilator technique, and will measure esophageal pressures to compare transpulmonary and respiratory system mechanics.

DETAILED DESCRIPTION:
This study will compare two different modes of mechanical ventilation: standard lung protective controlled mandatory ventilation and Adaptive Support Ventilation. The investigators will enroll adult patients with ARDS who are mechanically ventilated and admitted to intensive care units, capturing a population with respiratory failure and significant critical illness. Patient mechanics during each ventilation strategy will be compared before and after crossover.

After obtaining informed consent, the investigators will place an esophageal balloon which will be used for simultaneous measurements of airway pressures (Pao) and esophageal pressures (Pes), to estimate transpulmonary pressures (PL = Pao - Pes), while also measuring Flow and Volume. Use of esophageal balloon catheters is common practice in the ICUs, and standard of care at Beth Israel Deaconess Medical Center is to use these balloons in patients with ARDS. Both the respiratory therapy and physician staff are very comfortable with placement and use. The esophageal balloon will be left in place until extubation. If the balloon is dislodged or removed for clinical purposes, it will not be replaced solely for research purposes unless it occurs on the first day of study measurements.

Patients will then be randomized to be switched to ASV immediately or to be maintained on their current lung protective ventilation settings.

ELIGIBILITY:
Inclusion Criteria:

1. Patients ≥ 18 years of age
2. Receiving mechanical ventilation in an intensive care unit
3. ARDS, as defined by the Berlin definition:

   1. Hypoxemic respiratory failure with PaO2 / FiO2 ratio < 300 mmHg
   2. Bilateral alveolar/interstitial infiltrates on chest x-ray, with opacities not present for more than 7 days
   3. Respiratory failure not fully explained by cardiac failure or fluid overload
   4. Intubation on mechanical ventilation and receiving PEEP ≥ 5 cm H2O
4. Receiving mechanical ventilation from a Hamilton ventilator, on a controlled mode of ventilation.

Exclusion Criteria:

1. Clinical team refusal
2. Esophageal injury or contraindication precluding placement of the esophageal balloon

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2018-02-14 (Actual); Primary Completion 2020-11-02 (Actual); Study Completion 2021-01-31 (Actual)

PRIMARY OUTCOMES:
Tidal Volume | Day 1
  Lung tidal volume in both ventilation modes (mL)

SECONDARY OUTCOMES:
Driving Pressure (cmH20) | Day 1
  Driving pressure in both ventilation modes
Respiratory rate (BPM) | Day 1
  Respiratory Rate in both ventilation modes
Oxygenation (SpO2%) | Day 1
  Oxygenation (SpO2%) in both ventilation modes
CO2 clearance | Day 1
  CO2 clearance in both ventilation modes
Blood Gas pH | Day 1
  Blood Gas pH (units) in both ventilation modes
Blood Gas Partial Pressure of Oxygen | Day 1
  Partial pressure of oxygen (PaO2) (mm Hg) in both ventilation modes
Blood Gas Partial Pressure of Carbon Dioxide (PaCO2) (mm Hg) | Day 1
  Partial Pressure of Carbon Dioxide (PaCO2) (mm Hg) in both ventilation modes
Composite measure (lung protectiveness) - Asynchrony index | Day 1
  Asynchrony index
Composite measure (lung protectiveness) - Number of Adjustments | Day 1
  Number of Adjustments
Composite measure (lung protectiveness) - Time with tidal volumes under 6cc/kg | Day 1
  Time spent with tidal volumes less than or equal to 6cc/kg
Composite measure (lung protectiveness) - Driving pressures less than 15 | Day 1
  Time spent at or under Driving pressures less than 15
Composite measure (lung protectiveness) - Plateau Pressure <30 | Day 1
  Time spent at or under Plateau Pressure <30
Composite measure (lung protectiveness) - Oxygen saturation by pulse Oximetry (SpO2) >88% | Day 1
  Time spent at or under Oxygen saturation by pulse Oximetry (SpO2) >88%
Time to extubation | 30 Days
  Time to liberation from mechanical ventilation (days)
ICU length of stay | 90 Days
  Time to ICU discharge (days)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Talmor, MD, MPH, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided